CLINICAL TRIAL: NCT02418663
Title: Fluid Responsiveness in the Postoperative Patient: a Prospective Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Gabriele Baldini, MD, MSc, Assistant Professor, Assistant Professor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Not Applicable | Model: Single Group | Masking: Triple | Purpose: Screening
Other Study IDs: 14-452 SDR
Record Dates: First submitted 2015-03-16; First posted 2015-04-16 (Estimated); Last update posted 2015-05-15 (Estimated); Status verified 2015-04

CONDITIONS: Actual Impaired Fluid Volume
Keywords: fluid responsiveness; enhanced recovery program
MeSH Terms: interventions — Ringer's Lactate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Postoperative elective surgical patients (Other): Patients undergoing major elective thoracic and abdominal, the latter group including upper gastrointestinal, esophageal, and colorectal procedures. In this group FR will predicted by administering a fluid challenge of 250 ml of Lactated Ringer's solution and measuring SV with the ccNexfin
  Interventions: Drug: Fluid challenge (250 ml Lactated Ringer's solution)

INTERVENTIONS:
Drug: Fluid challenge (250 ml Lactated Ringer's solution) — When VE is prescribed to a patient, a fluid challenge of 250mL Lactated Ringer's solution will first be administered. The ccNexfin system will be used to predict FR (SV increases by at least 15% in response to a fluid challenge). The remaining amount of fluid ordered by the treating team will then be administered, and SV will again be measured.
  Additionally, a daily fluid challenge with 250mL of Lactated Ringer's will also be administered, with FR recorded as above
  Other Names: Lactated Ringer's Injection

SUMMARY:
The aim of this study is to determine the prevalence of Fluid Responsiveness (FR) (SV increases by at least 15% after Volume Expansion, VE) in postoperative patients admitted on a surgical ward after elective abdominal, thoracic and esophageal surgery

DETAILED DESCRIPTION:
Perioperative care

Preoperative Period

As per usual practice, the patient's staff surgeon will provide directives for preoperative fasting and fluid intake. These patients are encouraged to drink up to two hours before hospital admission, and also receive preoperative carbohydrate drinks the night before (100 grams), and the morning of surgery (50 grams) when indicated. Additionally, routine use of mechanical bowel preparation is avoided, and is prescribed only in selected cases. The patient's weight will be obtained upon arrival in the operating room.

Anesthetic and analgesic management

Anesthetic management and choice of postoperative analgesia will be as per usual care, at the discretion of the staff anesthesiologist in-charge of the case. An arterial line or central venous line may be inserted, and Goal Directed Fluid Therapy (GDFT) employed if deemed necessary.

Post-anesthesia Care Unit (PACU)

On arrival to the PACU, basic hemodynamic parameters, including heart rate (HR), blood pressure (BP), oxygen saturation, respiratory rate, temperature, and central venous pressure (CVP), if available, will be recorded according to standardized PACU protocol. A research assistant will then collect initial PACU values for these hemodynamic variables. Surgical time, estimated surgical blood loss, urine output, and intraoperative fluid and blood product administration will also be recorded. PACU care will be dictated by the treating staff anesthesiologists. Patients will be discharged from PACU according to standard institutional criteria.

Surgical floor

Postoperative care management, including the commencement of oral diet and fluid management, will be at the discretion of the surgical team. If required, VE (volume of the solution to be infused and type of the intravenous solution) will be decided case by case by the surgical team. The patient's weight will be obtained daily until hospital discharge. Patients will typically be discharged if afebrile, able to tolerate oral diet, pain is controlled (numeric rating scale (NRS) < 4), and they are able to ambulate.

Assessment of FR

A research assistant working in the department of Anesthesia will assess FR on two occasions:

1. When any VE is ordered by the treating team, either in PACU or on the surgical floor upon standard evaluation of hemodynamic parameters, urine output, surgical losses, and laboratory test abnormalities. FR will be assessed by measuring SV and Cardiac Output (CO) obtained by the ccNexfin system before 1 and 5 minute after VE. A patient will be considered a fluid responder if SV increases by at least 15% 1 minute after VE. A cut-off of 15% has been chosen as it represents the minimal clinical significant difference between two CO measurements obtained by thermodilution.
2. Upon arrival to the PACU, and every day before breakfast during the hospital stay. FR will be assessed by measuring SV and CO obtained by the ccNexfin system before and after 1 minute following 250 ml of Lactated Ringer's given as fluid challenge. A patient will be considered a fluid responder if SV increases by at least 15% after the fluid challenge.

Prediction of FR

A fluid challenge of 250 ml of Lactated Ringer's will be used to predict FR before the administration of any VE ordered by the treating team, either in PACU or on the surgical floor upon standard evaluation of hemodynamic parameters, urine output, surgical losses, and laboratory test abnormalities. A patient will be considered a fluid responder if SV increases by at least 15% 1 min after the end of a fluid challenge The utilization of fluid challenges has been shown to have high-accuracy (Receiver Operating Characteristic (ROC) curve of > 0.9) to predict FR in spontaneously breathing patients47. Furthermore, administration of fluid challenges to predict FR has already been described in several trials, including those with sick patient populations48 (ICU patients, patients undergoing major surgery, and patients with Ejection Fraction (EF) <40%).

Measurement of FR

1. Assessment of FR when VE is deemed necessary by the treating physician in PACU or on the surgical floor Prior to administration of a non-emergent fluid bolus (VE) ordered by the treating physician, nurses will additionally page the research assistant who will measure ccNexfin CO-Trek parameters as described earlier, and then administer a fluid challenge and measure FR. For simplicity, a single pager number will be used, and it will be affixed to the front of the chart of patients included in the study. A copy of the study protocol will also be given to nurses in the PACU and on the surgical floors for perusal.

   The need for VE will be evaluated by the anesthetist in charge in PACU, or by the surgical team on the surgical ward. Hemodynamic variables triggering fluid administration will be decided based on standard evaluation of hemodynamic parameters, urine output, surgical losses, and laboratory test abnormalities. The type and amount of intravenous solution to be used will be decided by the anesthetist in charge or by the surgical team.

   Before VE, hemodynamic variables including HR and BP will be measured by the research assistant. CVP will me measured in PACU if patients receive a central venous catheter. Then, the ccNexfin system will be applied in a standardized fashion according to manufacturer recommendations: an appropriately sized finger cuff will be selected and placed around the patient's middle finger. The wrist unit and heart reference sensor (HRS) will then be placed around the patient's wrist and ring finger respectively. The system will be zeroed, and the sensor end of the HRS will be placed at the level of the patient's heart, which allows for compensation for hydrostatic pressure differences between the finger and the heart. The ccNexfin will then calculate and display the values for an initial post-operative CO, Cardiac Index (CI), and SV. One and 5 minutes after the end of the VE, the same hemodynamic parameters will be measured. Should any further bolus of fluid be administered, FR and basic hemodynamic variables will be measured as above, upon administration of VE as ordered by the treating team.
2. Prediction of FR before the administration of any VE ordered by the treating team

   A fluid challenge of 250 ml of Lactated Ringer's solution (Baxter, Lactated Ringer's Injection, USP, 1000 mL VIAFLEX Plastic Container) will be administered over 5 minutes by the research assistant before VE. One and 5 minutes following the end of the fluid challenge, basic hemodynamic values (as described above), as well as CO, CI, and SV obtained from the ccNexfin system, will again be recorded. An increase of SV by at least 15% 1 minute after the end of the fluid challenge will be considered clinically significant. Upon termination of a fluid challenge, the decision on weather to proceed with VE will be taken by the treating physician based only on standard signs and measures of hypovolemia and not on any of the ccNexfin SV and CO measurements obtained during the fluid challenge. The proportion of patients identified as fluid responsive after VE will be compared with the proportion of patients responding to the fluid challenge.

   The research assistant will be available to measure FR from 6.30 AM to 7.30 PM every day during patient hospitalization. For patient safety, the research assistant must arrive at the bedside within ten minutes of being paged, in order to measure FR before VE. Intravenous fluids will be administered without measuring CO and administering a fluid challenge if:
   1. the research assistant will not be able to arrive at the bedside within ten minutes;
   2. the treating physician considers immediate administration of intravenous fluids necessary.

   CO measurements will not be taken before administering blood products. Blood product administration (erythrocytes, platelets, fresh frozen plasma, or cryoprecipitate) will also be at the discretion of the staff anesthetist (in PACU) or at the discretion of the surgical team (surgical ward).
3. Daily assessment of FR

After surgery in PACU, and daily (before breakfast) for the duration of the patient's hospital stay a research assistant will administer a fluid challenge. As described above, CO, CI, and SV will be measured by the research assistant using the ccNexfin system, to assess for FR. A fluid challenge of 250 ml of Lactated Ringer's solution (Baxter, Lactated Ringer's Injection, USP, 1000 mL VIAFLEX Plastic Container) will then be administered over 5 minutes. One and 5 minutes following fluid challenge completion, basic hemodynamic values (as described above), as well as CO, CI, and SV obtained from the ccNexfin system, will again be recorded. An increase of SV by at least 15% 1 minute after the end of the fluid challenge will be considered clinically significant.

Daily assessment of FR, regardless of whether patients will receive intravenous fluids, will determine if FR is associated with an increased risk of complications and/or prolonged hospital stay.

All ccNexfin values obtained before and after VE and any fluid challenge will be blinded to the treating anesthetist, the surgical team and the nursing team.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing major elective thoracic and abdominal surgeries, the latter group including upper gastrointestinal, esophageal, and colorectal procedures,
* Patients treated with surgery-specific enhanced recovery programs (ERPs), implemented in 2010 at the Montreal General Hospital for colorectal surgery, and subsequently developed at the same institution for thoracic surgery

Exclusion Criteria:

* Age <18 years
* Emergency surgery
* Patients who do not understand, read or communicate in either French or English
* Chronic kidney disease
* Congestive heart failure
* Severe aortic stenosis
* Patients not in sinus rhythm
* Patients requiring fluid restriction for any reason
* Known peripheral vascular disease or Raynaud's phenomenon
* Septic patients
* Acute circulatory shock

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 245 (Estimated)
Dates: Start 2015-06; Primary Completion 2017-04 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
FR assessed by the ccNexfin system, anytime VE is ordered by the treating physician | For the entire duration of hospital stay (an average of 3 days for patients undergoing colorectal surgery, 4 days for patients undergoing thoracic surgery, and 6 days for patients undergoing esophageal surgery)
  FR (SV increases by ≥ 15% ) FR will be measured 1 minute after the completion of VE

SECONDARY OUTCOMES:
Prediction of FR | For the entire duration of hospital stay (an average of 3 days for patients undergoing colorectal surgery, 4 days for patients undergoing thoracic surgery, and 6 days for patients undergoing esophageal surgery)
  The probability of being fluid responsive after VE will be tested before initiating VE by administering a fluid challenge of 250 ml of Lactated Ringer's. The patient will be considered fluid responder to the fluid challenge if SV increases by ≥ 15% 1 minute after the infusion
FR assessed by the ccNexfin system, at the arrival in PACU and daily on the surgical floor | At the arrival in PACU and daily for the entire duration of hospital stay (an average of 3 days for patients undergoing colorectal surgery, 4 days for patients undergoing thoracic surgery, and 6 days for patients undergoing esophageal surgery)
  FR (SV increases by ≥ 15% ) FR will be measured 1 and 5 minutes after the completion of the fluid challenge of 250 ml of Lactated Ringer's.
Dynamic Arterial Elastance (absolute number), anytime VE is ordered by the treating physician | Before the fluid challenge, for the entire duration of hospital stay (an average of 3 days for patients undergoing colorectal surgery, 4 days for patients undergoing thoracic surgery, and 6 days for patients undergoing esophageal surgery)
  Ratio between Pulse Pressure Variation (PPV,%) and Stroke Volume Variation (SVV,%)
Heart rate (beat per minute) | At the arrival in PACU and daily for the entire duration of hospital stay (an average of 3 days for patients undergoing colorectal surgery, 4 days for patients undergoing thoracic surgery, and 6 days for patients undergoing esophageal surgery)
Arterial Blood Pressure (mmHg) | At the arrival in PACU and daily for the entire duration of hospital stay (an average of 3 days for patients undergoing colorectal surgery, 4 days for patients undergoing thoracic surgery, and 6 days for patients undergoing esophageal surgery)
Central Venous Pressure (CVP)(mmHg) | At the arrival in PACU, if available
Urine output | At the arrival in PACU,and daily for the entire duration of hospital stay (an average of 3 days for patients undergoing colorectal surgery, 4 days for patients undergoing thoracic surgery, and 6 days for patients undergoing esophageal surgery)
Respiratory Rate (breaths per minutes) | At the arrival in PACU,and daily for the entire duration of hospital stay (an average of 3 days for patients undergoing colorectal surgery, 4 days for patients undergoing thoracic surgery, and 6 days for patients undergoing esophageal surgery)
Peripheral Oxygen Saturation (%) | At the arrival in PACU,and daily for the entire duration of hospital stay (an average of 3 days for patients undergoing colorectal surgery, 4 days for patients undergoing thoracic surgery, and 6 days for patients undergoing esophageal surgery)
Amount of perioperative intravenous fluids administered | At the arrival in PACU and daily for the entire duration of hospital stay (an average of 3 days for patients undergoing colorectal surgery, 4 days for patients undergoing thoracic surgery, and 6 days for patients undergoing esophageal surgery)
24 hour postoperative weight gain | Daily for the entire duration of hospital stay (an average of 3 days for patients undergoing colorectal surgery, 4 days for patients undergoing thoracic surgery, and 6 days for patients undergoing esophageal surgery)
Quality of recovery measured by the Quality of Recovery Score | Daily for the entire duration of hospital stay (an average of 3 days for patients undergoing colorectal surgery, 4 days for patients undergoing thoracic surgery, and 6 days for patients undergoing esophageal surgery)
  Score 0-18
Number of patients with at least one postoperative complication | Daily for the entire duration of hospital stay (an average of 3 days for patients undergoing colorectal surgery, 4 days for patients undergoing thoracic surgery, and 6 days for patients undergoing esophageal surgery)
  Postoperative complications will be defined a priori and classified based on Clavien Classification
Number of postoperative complications | Daily for the entire duration of hospital stay (an average of 3 days for patients undergoing colorectal surgery, 4 days for patients undergoing thoracic surgery, and 6 days for patients undergoing esophageal surgery)
  Postoperative complications will be defined a priori and classified based on Clavien Classification
Type of postoperative complication | Daily for the entire duration of hospital stay (an average of 3 days for patients undergoing colorectal surgery, 4 days for patients undergoing thoracic surgery, and 6 days for patients undergoing esophageal surgery)
  Postoperative complications will be defined a priori and classified based on Clavien Classification
Readiness to be discharged | Daily for the entire duration of hospital stay (an average of 3 days for patients undergoing colorectal surgery, 4 days for patients undergoing thoracic surgery, and 6 days for patients undergoing esophageal surgery)
  Elapsed time (days) between surgical admission (same day of surgery) and the achievement of hospital discharge criteria
Length of hospital stay | Daily for the entire duration of hospital stay (an average of 3 days for patients undergoing colorectal surgery, 4 days for patients undergoing thoracic surgery, and 6 days for patients undergoing esophageal surgery)
  Elapsed time (days) between surgical admission (same day of surgery) and primary hospital discharge. The day of surgery is count as postoperative day 0
30 days readmission rates | 30 days after primary hospital discharge following surgery

OTHER OUTCOMES:
Incidence of arterial hypotension, defined as Systolic Blood Pressure less than 90 mmHg or less than 20% of the baseline value | At the Arrival in PACU and daily for the entire duration of hospital stay (an average of 3 days for patients undergoing colorectal surgery, 4 days for patients undergoing thoracic surgery, and 6 days for patients undergoing esophageal surgery)
Estimated surgical blood loss | At the end of surgery
Amount of volume expansion administered by the treating team | At the Arrival in PACU and daily for the entire duration of hospital stay (an average of 3 days for patients undergoing colorectal surgery, 4 days for patients undergoing thoracic surgery, and 6 days for patients undergoing esophageal surgery)
Indications justifying volume expansion | At the Arrival in PACU and daily for the entire duration of hospital stay (an average of 3 days for patients undergoing colorectal surgery, 4 days for patients undergoing thoracic surgery, and 6 days for patients undergoing esophageal surgery)
  Any clinical indication or laboratory abnormality triggering volume expansion
Number of patients (reported as percentage) requiring intraoperative and post operative Vasopressors in PACU | During PACU stay, an average of 3-6 h depending on the type of surgery
Intraoperative and postoperative urinary output | During surgery, in PACU and daily for the entire duration of hospital stay (an average of 3 days for patients undergoing colorectal surgery, 4 days for patients undergoing thoracic surgery, and 6 days for patients undergoing esophageal surgery)
Daily postoperative pain: numerical rating scale (NRS), at rest, on coughing and ambulating | Daily for the entire duration of hospital stay (an average of 3 days for patients undergoing colorectal surgery, 4 days for patients undergoing thoracic surgery, and 6 days for patients undergoing esophageal surgery)

CONTACTS AND LOCATIONS:
Overall Officials: Gabriele Baldini, MD, MSc, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre

REFERENCES:
- [Background] Myles PS, Hunt JO, Nightingale CE, Fletcher H, Beh T, Tanil D, Nagy A, Rubinstein A, Ponsford JL. Development and psychometric testing of a quality of recovery score after general anesthesia and surgery in adults. Anesth Analg. 1999 Jan;88(1):83-90. doi: 10.1097/00000539-199901000-00016. PMID 9895071
- [Background] Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83. doi: 10.1016/0021-9681(87)90171-8. PMID 3558716